CLINICAL TRIAL: NCT00744315
Title: Induced Angiogenesis by Genic Therapy With VEGF165 in Advanced Ischemic Cardiomyopathy - Historical Controlled Trial
Brief Title: Induced Angiogenesis by Genic Therapy in Advanced Ischemic Cardiomyopathy
Acronym: THEANGIOGEN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Imarilde Giusti, Institute of Cardiology of Rio Grande do Sul/FUC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP3549
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-07

CONDITIONS: Ischemic Cardiopathy
Keywords: myocardial revascularization; myocardial ischemia; genetics, medical; Angiogenesis Inducing Agents
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Controlled
  Interventions: Procedure: Mini-thoracotomy for intramyocardial injection of VEGF165

INTERVENTIONS:
Procedure: Mini-thoracotomy for intramyocardial injection of VEGF165 — Patients with previous diagnosis of ischemic cardiopathy were included. The patient must accept and agree to be subject of clinical observation with current optimal treatment for at least 6 months. Following to that, subject undergoes intervention, in addition to consultation and assessments. Surgical technique -Ten injections VEGF165 will be made through a 25F butterfly needle in any ischemic territory where previously identified through scintigraphy. Dosis: 2.000 mg of VEGF165 in 5ml of saline solution. After the procedure, the patients will be kept in a recovery room for about 24hs and in the hospital until full clinical recovery.

SUMMARY:
Human Vascular Endothelial Grown Factor 165 (hVEGF165) administration is promising therapy induces a new vessels, arterioles and capillaries in regions whose revascularization surgery is not possible by direct or by percutaneous angioplasty. This study aims to evaluate the clinical effects and safety of gene therapy with hVEGF165 in patients with advanced coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis coronary artery disease and symptomatic, despite optimal pharmacologic therapy
* Left ventricular dysfunction - left ventricular ejection fraction between 60% and 25% by echocardiogram
* Non-conventional revascularization, as seen by cineangiocardiography, attested by interventional cardiologist and cardiac surgeon
* Age below 75 years
* Absence of neoplasm

Exclusion Criteria:

* No

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Clinical finds | eighteen months

CONTACTS AND LOCATIONS:
Overall Officials: Renato AK Kalil, MD, PhD, Study Director — Scientific Direction - Institute of Cardiology of Rio Grande do Sul / FUC
Locations (1):
- Institute of Cardiology of Rio Grande do Sul / FUC, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Giusti II, Rodrigues CG, Salles FB, Sant'Anna RT, Eibel B, Han SW, Ludwig E, Grossman G, Prates PR, Sant'Anna JR, Filho GF, Markoski MM, Nesralla IA, Nardi NB, Kalil RA. High doses of vascular endothelial growth factor 165 safely, but transiently, improve myocardial perfusion in no-option ischemic disease. Hum Gene Ther Methods. 2013 Oct;24(5):298-306. doi: 10.1089/hgtb.2012.221. PMID 23944648